CLINICAL TRIAL: NCT03793907
Title: Feasibility of Strength Training and Impact on Pain and Quality of Life in Patients With Multiple Myeloma
Brief Title: Strength Training in Improving Pain and Quality of Life in Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: i 70118; i 70118 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-12-28; First posted 2019-01-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 2 (walking program) (Active Comparator): Patients receive a Fitbit to track their physical activity, and complete an unsupervised walking program daily at home, increasing physical activity stepwise weekly, for 6 months.
  Interventions: Device: FitBit; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: STEPS to Enhance Physical Activity
- Cohort 1 (strength training) (Experimental): Patients receive a Fitbit to track their physical activity, and complete an in-person personalized and supervised full-body strength training program over 1 hour BID up to 52 sessions for 6 months.
  Interventions: Device: FitBit; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Device: FitBit — Wear Fitbit
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Complete strength training
  Other Names: Strength Training
  Arms: Cohort 1 (strength training)
Behavioral: STEPS to Enhance Physical Activity — Complete a walking program
  Other Names: STEPS; STEPS Intervention; STEPS to Enhance Physical Activity (STEPS)
  Arms: Cohort 2 (walking program)

SUMMARY:
This trial studies how well strength training works in improving bone health, pain, and quality of life in patients with multiple myeloma. Weekly physical activity may improve bone recovery, reduce pain, and increase quality of life in patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. To assess the feasibility of a 6 month, twice weekly supervised strength training intervention in patients with multiple myeloma. (Cohort 1)
* II. To assess the feasibility of a 6 month behavioral intervention to prompt an increase in weekly physical activity in patient with multiple myeloma. (Cohort 2)

SECONDARY OBJECTIVES:

I. To assess the adherence rate of patients during a 6 month intervention program.

II. To assess the eligibility and recruitment rate for the trial among patients with multiple myeloma.

EXPLORATORY OBJECTIVES:

I. Comparison of disease activity parameters, physical activity level, clinical symptoms, medication, psycho-oncological parameters before, during and after intervention.

II. Determine factors that may influence a persons' willingness to participate in the trial.

III. Investigate "immune fitness" by frequencies and function of immune cell subsets in peripheral blood.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHRT 1 (STRENGTH TRAINING): Patients receive a Fitbit to track their physical activity, and complete an in-person personalized and supervised full-body strength training program over 1 hour twice weekly (BID) up to 52 sessions for 6 months.

COHORT 2 (BEHAVIORAL INTERVENTION): Patients receive a Fitbit to track their physical activity, and complete an unsupervised walking program daily at home, increasing physical activity stepwise weekly, for 6 months.

After completion of study, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Have a diagnosis of multiple myeloma
* Show no signs of comorbidities, myeloma symptoms, or treatment side effects that would put them in danger when participating in the study according to the physician's discretion
* Are able to understand and follow assessment and training procedures
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Current and symptomatic pathological fracture(s) or severely advanced instability of the musculo-skeletal system
* Acute bone instability as assessed by whole body low-dose computed tomography and evaluated by an experienced neuro- and spine surgeon
* Major comorbidities that would cause danger to the patient when participating in the study. Examples are cardiac or pulmonary and infectious diseases that would have a risk of progression if the patient took part in the study
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to take part in study intervention (comorbidities, myeloma symptoms, treatment side effects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Feasibility rate | At 6 months
  Will be defined as the proportion of enrolled patients who are still on study at the end of 6 months. Analysis will be done via computing a two-sided 95% confidence interval for the true proportion using Clopper-Pearson method.

SECONDARY OUTCOMES:
Adherence rate (Cohort 1) | At 6 months
  Will be defined as the proportion of patients remaining on study at 6 months who complete >= 80% of the intervention activities. Analysis will be done via computing a two-sided 95% confidence interval for the true proportion using Clopper-Pearson method.
Adherence rate (Cohort 2) | At 6 months
  Will be defined as the proportion of patients whose average daily step counts each week are at or above their goal for that week at least 20/26 weeks, or 80% of the weeks.

OTHER OUTCOMES:
Differences in lab parameters | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Clinical performance | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Physical activity level | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Pain | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Polyneuropathy | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Opioid and other drug consumption | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Psycho-oncological parameters | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Fatigue | Before, during and after strength training program
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments.
Reasons why patients do not participate in the trial | Before and after strength training program up to 1 year
  Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments. This will be assessed by analysis of the screening questionnaires and the checklist.
"Immune fitness" frequencies and function of immune cell subsets | Before and after strength training program up to 1 year
  Will be measured in peripheral blood. Comparison of parameters before and after intervention for the exploratory endpoints will proceed using two-sided paired t-tests for significance at the alpha = 0.05 level for continuous measures, and sign- tests for ordinal outcomes. Multiple testing corrections will make use of Bonferroni adjustments. This will be assessed by analysis of the screening questionnaires and the checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hillengass, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States